CLINICAL TRIAL: NCT05833308
Title: Association Between Fibrinogen-to-albumin Ratio and Delirium After Deep Brain Stimulation Surgery in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wen-bin Lu, MD, Principal Investigator, Changhai Hospital
Other Study IDs: POD-FAR
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease; Deep Brain Stimulation; Postoperative Delirium
Keywords: postoperative delirium; fibrinogen-to-albumin ratio
MeSH Terms: conditions — Parkinson Disease; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: Patients who were determined to have incident postoperative delirium by a positive confusion assessment method (CAM) questionnaire after operation were defined as the POD group.
- Non-POD group: Patients who did not suffer from delirium after surgery consisted of the Non-POD group.

SUMMARY:
Postoperative delirium (POD) remains one of the most common neuropsychiatric complications after deep brain stimulation (DBS) surgery. The fibrinogen-to-albumin ratio (FAR) has been shown to significantly correlate with prognosis of many diseases associated with inflammation, but the relationship between FAR and POD is unclear. The investigators aimed to investigate the association between POD and FAR in Parkinson's disease (PD) patients receiving DBS surgery. For this aim, the present study was conducted to provide a new method for the early recognition and perioperative management of delirium after DBS surgery in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 55 years old
* American Society of Anesthesiologists (ASA) physical status I-III
* Bilateral subthalamic nucleus deep brain stimulation surgery

Exclusion Criteria:

* Preoperative delirium
* Missing preoperative laboratory parameters on fibrinogen or albumin
* Persistent infectious diseases
* Coagulopathy and autoimmune-illness or malignancies

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease were scheduled to undergo elective subthalamic nucleus deep brain stimulation surgery for the first time under total intravenous anesthesia. Delirium was evaluated at the preoperative visit, then twice daily for 3 days following surgery. Cognition assessment was conducted at preoperative visit, 24 h after surgery and 72 h after surgery. Delirium assessments were performed before 10 AM and after 5 PM in the ward. The CAM questionnaire and cognition assessment method for MMSE were performed by the qualified doctor who trained with CAM and MMSE training manual.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
CAM score | Before surgery
  Positive CAM score means that patient developed delirium after surgery. While negative CAM score means that patient did not suffer from delirium after surgery.
CAM score | Postoperative day 1
  Positive CAM score means that patient developed delirium after surgery. While negative CAM score means that patient did not suffer from delirium after surgery.
CAM score | Postoperative day 2
  Positive CAM score means that patient developed delirium after surgery. While negative CAM score means that patient did not suffer from delirium after surgery.
CAM score | Postoperative day 3
  Positive CAM score means that patient developed delirium after surgery. While negative CAM score means that patient did not suffer from delirium after surgery.

SECONDARY OUTCOMES:
Mini-mental State Examination (MMSE) score | Before surgery
  MMSE score ranges from 0 to 30 and higher score means better cognitive function.
MMSE score | Postoperative 24 hour
  MMSE score ranges from 0 to 30 and higher score means better cognitive function.
MMSE score | postoperative 72 hour
  MMSE score ranges from 0 to 30 and higher score means better cognitive function.
The level of fibrinogen-to-albumin ratio (FAR) in peripheral blood. | Before surgery
  The FAR was calculated as fibrinogen / albumin.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China